CLINICAL TRIAL: NCT04183933
Title: The Effect of Different Exercise Training on Balance and Functional Status in Individuals With Osteoarthritis'
Brief Title: The Effect of Exercise Training on Balance and Functional Status in Individuals With Osteoarthritis'
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Berkiye Kırmızıgil, Director, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETK00-2019-0206
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Osteo Arthritis Knee; Balance
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Exercise Group (Active Comparator): Pilates exercises will given for 6 weeks, 3 days in a week.
  Interventions: Other: Pilates Exercise
- Combined Exercise group (Active Comparator): Combined exercises will given for 6 weeks, 3 days in a week.
  Interventions: Other: Combined Exercise

INTERVENTIONS:
Other: Pilates Exercise — Pilates exercises will be given for 6 weeks, 3 days in a week.
  Arms: Pilates Exercise Group
Other: Combined Exercise — Combined exercise will be given for 6 weeks, 3 days in a week.
  Arms: Combined Exercise group

SUMMARY:
The aim of this study was to evaluate and compare the effects of Clinical Pilates Exercise Training and Combined Exercise Training on balance and functional status in individuals with knee Osteoarthritis (OA).

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with knee osteoarthritis II-III level according to the results of radiological evaluation by Kellgren and Lawrence

  * Individuals aged between 40 and 70 years
  * Individuals who have pain in his/her either of the knees in 3 month period and who have a VAS score of 3 or more
  * Individuals who can walk 10 meters independently (with or without ancillary device)

Exclusion Criteria:

* Individuals with Body Mass Index 35 and above
* Individuals with a history of surgery or injury involving the lower limb within the last 1 year (knee / hip endoprosthesis, post-fracture surgery, menisectomy, etc.)
* Individuals who received hyaluronic acid or corticosteroid injections in the last year
* People with severe eyesight, hearing disabilities Individuals with neurological deficit or disorder
* Individuals with regular exercise habits in the last 6 months
* Individuals with inflammatory rheumatic diseases.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-01-24 (Estimated); Study Completion 2020-02-10 (Estimated)

PRIMARY OUTCOMES:
Fullerton Advanced Balance Scale (FAB-T) | Change will be assessed from the baseline at 1 week and 6th week
  It is a test that determines the functional balance state of individuals. The test has 10 parameters. These are: feet adjacent and eyes closed standing, reaching out forward to reach a shoulder-length object, 360 degrees of turning in right and left directions, stepping and passing over a 15.24 cm-long stair, tandem march, standing on one leg, eyes closed staying on the foam, double feet bounce, walking with head turning, reactive postural control. In this scale, which is scored between 0-40, a score between 0 and 4 is given for each item.

SECONDARY OUTCOMES:
Berg Balance Test | Evaluation will be applied on the first day and after 6 weeks
  is a routine test used in daily life, consisting of evaluation of 14 activities, requiring both dynamic and static balance. If the total score is between 0 and 20, there is a high risk of falling, between 21 and 40 there is a moderate risk of falling, between 41-56 there is a low risk of falling.
The Timed Up & Go (TUG) Test | Change will be assessed from the baseline at 1 week and 6th week
  TUG is a frequently used balance test to assess the functional mobility of individuals. It was developed by Podsiadlo and Richardson in 1991. Test measures the speed during many functional maneuvers such as standing up, walking, turning and sitting. In the test, the person is asked to get up from the chair, to walk for 3 meters with his/her own normal speed, to walk back and to sit on the chair and the time is recorded in seconds (sec). A shorter time indicates better balance and mobility. The starting position should be standardized. It is performed 3 times and the average value is recorded
Single Leg Stance Test on Hard Ground | Change will be assessed from the baseline at 1 week and 6th week
  the patient is asked to flex the knee with eyes open, hands on the hips, feet naked, and the hip in neutral position. The time is started as soon as the foot is removed from the ground and recorded in seconds. The patient is asked to stand on one foot until the arms move or until the foot is dropped on the floor or until the time reaches 60 sec. For each foot, 3 attempts are made and the average time for each foot is recorded. Rest is allowed between attempts
Single Leg Stance Test on Foam Ground | Change will be assessed from the baseline at 1 week and 6th week
  Eyes open, hands on the hips, feet naked, hip in neutral position on the foam, participant is required to flex a knee. The patient is asked to stand on one foot until the arms move or until the foot is dropped on the floor or until the time reaches 60 sec. For each foot, 3 attempts are made and the average time for each foot is recorded. Rest is allowed between attempts.
Push and Release Test | Change will be assessed from the baseline at 1 week and 6th week
  While the patient is in the standing position with the eyes open, the physiotherapist stands behind the person and places his/her hand on the person's scapula and participant leans backwards to push the hand of the physiotherapist.
  The physiotherapist flexes the elbows to allow back movement of the body and supports the person's weight with his/her hands. When a person's shoulders and hips are in a fixed position just behind the heels, the physiotherapist suddenly raises participant's hands.
30 Seconds Sit and Stand Up Test | Change will be assessed from the baseline at 1 week and 6th week
  For proximal muscle strength of the lower extremity and endurance, this test is valid and reliable for adults. In his/ her starting position, the person sits on an armless armchair with his back straight, arms crossed in front of the chest and feet on the ground. With the starting of the measument, the person takes the sitting position from a full standing position and the exact numbers of standing uıp within 30 seconds are recorded. Less than 10 repetitions in 30 seconds show lower extremity muscle weakness
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index | Change will be assessed from the baseline at 1 week and 6th week
  consists of 24 questions and is divided into 3 subgroups. WOMAC subgroups consisted of 5 pain-related questions, 2 stiffness-related questions, 17 physical function-related problems. In WOMAC assessment, each question is between 0-4 points. Subgroups are evaluated among themselves. According to this, the subgroup of pain is 0-20 points, the stiffness / rigidity is 0-8 points and the physical function subgroup is 0-68 points. During the evaluation of pain, the severity of pain in the last 24 hours is questioned. For stiffness / rigidity sub-parameters, first; the feeling of stiffness is defined and the joint stiffness felt within the last 24 hours in the evaluated joint is questioned. For physical function score, 17 activities that is being challenging for the participant due to arthralgia in the joint is being questioned.
Four Step Square Test | Change will be assessed from the baseline at 1 week and 6th week
  4 squares are formed perpendicular to each other on a flat surface. All squares are numbered. At the beginning of the test, the patient standing in frame 1 with her face directed to frame 2 is instructed to take steps in succession (2-3-4-1-4-3-2-1) to each frame as quickly as possible without touching it.
  Individuals are said to be in contact with the ground with both feet in each frame (requiring the patient to step forward, backward, right and left sides). The completion time is recorded as a score. Two scores are measured, the best one is taken. The time is started when the first leg touches the ground on the second frame and ends with the last leg touching the ground on the first frame.

CONTACTS AND LOCATIONS:
Overall Officials: Gozde Iyigun, Asst. Prof, Principal Investigator — Eastern Mediterranean University; Sevim Oksuz, Asst. Prof, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided